CLINICAL TRIAL: NCT03801473
Title: Comparison of Robot-Assisted Gait Training and Conventional Therapy in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tugba Ozsoy
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: rehabilitation; robot assisted gait training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Initial assessments will be performed by first clinician (EA). Then, patients will be randomly grouped. The outcome assessor, second clinician (TOU) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot assisted training (RAT) (Experimental): RoboGait which is an automated locomotor therapy system was used for treating RAT group. The system composed of a robotic lower extremity orthosis, adjustable dynamic gait support, synchronized treadmill and biofeedback utilities
  Interventions: Other: robot assisted gait therapy
- conventional training (CT) (Active Comparator): Participants in CT group had physiotherapist assisted walking exercises on the parallel bars and on the ground with aids/cane, tripod or walker.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: robot assisted gait therapy — The Robogait is a fixed lower body hip-knee exoskeleton. The user's weight is supported by a combination of an overhead attached harness and the support from the exoskeleton.
  Arms: robot assisted training (RAT)
Other: Conventional rehabilitation — Conventional rehabilitation program. Exercise and walking education is performed by the physiotherapists.
  Arms: conventional training (CT)

SUMMARY:
The aim of this study is to compare conventional neurorehabilitation with robot-assisted gait training program in terms of fatigue, anxiety, depression and quality of life.

DETAILED DESCRIPTION:
Gait disturbances are common in Multiple Sclerosis (MS) patients. Nowadays, gait training with robot assisted technology is used for rehabilitation. In several studies conventional rehabilitation was compared with robot assisted rehabilitation program, and they found no superior effects of robot assisted walking program. In this study we aimed to compare these modalities in terms of fatigue, anxiety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old Multiple Sclerosis patients
* EDSS score: 5.5-7.5
* Being oriented and cooperated
* Mini-mental score ≥24/30

Exclusion Criteria:

* Modified Ashworth >3 in lower extremity muscles
* Cognitive impairment
* Botox injection within last 6-months
* Having another neurological disease
* Pregnancy or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefeber N, Swinnen E, Kerckhofs E. The immediate effects of robot-assistance on energy consumption and cardiorespiratory load during walking compared to walking without robot-assistance: a systematic review. Disabil Rehabil Assist Technol. 2017 Oct;12(7):657-671. doi: 10.1080/17483107.2016.1235620. Epub 2016 Oct 20. PMID 27762641
- [Background] Straudi S, Manfredini F, Lamberti N, Zamboni P, Bernardi F, Marchetti G, Pinton P, Bonora M, Secchiero P, Tisato V, Volpato S, Basaglia N. The effectiveness of Robot-Assisted Gait Training versus conventional therapy on mobility in severely disabled progressIve MultiplE sclerosis patients (RAGTIME): study protocol for a randomized controlled trial. Trials. 2017 Feb 27;18(1):88. doi: 10.1186/s13063-017-1838-2. PMID 28241776
- [Background] Gandolfi M, Geroin C, Picelli A, Munari D, Waldner A, Tamburin S, Marchioretto F, Smania N. Robot-assisted vs. sensory integration training in treating gait and balance dysfunctions in patients with multiple sclerosis: a randomized controlled trial. Front Hum Neurosci. 2014 May 22;8:318. doi: 10.3389/fnhum.2014.00318. eCollection 2014. PMID 24904361
- [Derived] Ozsoy-Unubol T, Ata E, Cavlak M, Demir S, Candan Z, Yilmaz F. Effects of Robot-Assisted Gait Training in Patients With Multiple Sclerosis: A Single-Blinded Randomized Controlled Study. Am J Phys Med Rehabil. 2022 Aug 1;101(8):768-774. doi: 10.1097/PHM.0000000000001913. Epub 2021 Oct 21. PMID 34686632

RESULTS

PARTICIPANT FLOW:
Groups:
- Robot Assisted Gait: robot assisted gait therapy: The Robogait is a fixed lower body hip-knee exoskeleton. The user's weight is supported by a combination of an overhead attached harness and the support from the exoskeleton.
Period: Overall Study
Arm/Group | Robot Assisted Gait | Conventional Rehabilitation
Started | 21 | 21
Completed | 18 | 19
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT) | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9.2) | 44.7 (8.4) | 44.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease duration [Mean (Standard Deviation); unit: years] | 14.1 (5.9) | 13.4 (6.2) | 13.7 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Score
Description: Patient-reported outcome measure which is composed of 9 items and evaluates the severity of fatigue. The items are scored on a 7-point scale with 1=strongly disagree and 7=strongly agree. The minimum score is 9 and maximum possible score is 63. FSS score is calculated as total score/9. Higher score reflects greater fatigue severity.
Time Frame: baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 5.5 [4.11 to 7] | 6 [4.11 to 7]

2. Primary Outcome: Fatigue Severity Score
Description: as for outcome 1
Time Frame: after treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 4.4 [3.00 to 6.44] | 5.8 [3.89 to 6.89]

3. Primary Outcome: Fatigue Severity Score
Description: as for outcome 1
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 5.5 [3.33 to 7] | 5.7 [4 to 7]

4. Primary Outcome: Hospital Anxiety Depression Scale-Depression Subscale (HADS-D)
Description: Hospital Anxiety Depression Scale (HADS) s a 14 item questionnaire which consists two sub-scale evaluating anxiety (HADS-A) and depression (HADS-D).
  HADS-D sub-scale has seven items and each item is scored on a scale of 0 to 3. Total score ranged from 0 to 21. Higher scores reflects more severe depression.
Time Frame: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 8.5 [0 to 12] | 10 [1 to 15]

5. Primary Outcome: Hospital Anxiety Depression Scale- Depression Subscale (HADS-D)
Description: as for outcome 4
Time Frame: After treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 5.5 [0 to 12] | 9 [1 to 15]

6. Primary Outcome: Hospital Anxiety Depression Scale- Depression Subscale (HADS-D)
Description: as for outcome 4
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 6.5 [0 to 13] | 9 [1 to 16]

7. Primary Outcome: Hospital Anxiety Depression Scale- Anxiety Subscale (HADS-A)
Description: Hospital Anxiety Depression Scale (HADS) s a 14 item questionnaire which consists two sub-scale evaluating anxiety (HADS-A) and depression (HADS-D).
  HADS-A sub-scale has seven items and each item is scored on a scale of 0 to 3. Total sub-scale score ranged from 0 to 21. Higher score mean a worse outcome.
Time Frame: baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 7.5 [3 to 13] | 8 [3 to 16]

8. Primary Outcome: Hospital Anxiety Depression Scale-Anxiety Subscale (HADS-A)
Description: as for outcome 7
Time Frame: After treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 5 [1 to 17] | 8 [3 to 15]

9. Primary Outcome: Hospital Anxiety Depression Scale-Anxiety Subscale (HADS-A)
Description: as for outcome 7
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 5 [2 to 15] | 8 [2 to 16]

10. Secondary Outcome: Multiple Sclerosis Quality of Life-54 (MSQOL-54)-Physical Health
Description: The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items.
  This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function.
  The summary scores are the physical health composite summary and the mental health composite summary.
  Each composite summary scored 0-100. Higher values indicate better QoL.
Time Frame: baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 28.5 [14.4 to 65.1] | 29.9 [10.8 to 63.1]

11. Secondary Outcome: Multiple Sclerosis Quality of Life-54 (MSQOL-54)-Physical Health
Description: as for outcome 10
Time Frame: after treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 34.2 [16.7 to 70.8] | 33.7 [16.2 to 73.4]

12. Secondary Outcome: Multiple Sclerosis Quality of Life-54 (MSQOL-54)- Physical Health
Description: as for outcome 10
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 32.9 [17.1 to 70.8] | 29.1 [16.2 to 65.1]

13. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: The EDSS assesses the disability status of MS patients on a scale range from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Time Frame: baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
units on a scale | 6.5 [5.5 to 7] | 6 [5.5 to 7]

14. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: as for outcome 13
Time Frame: after treatment (4th week)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
units on a scale | 6 [5.5 to 7] | 6 [5.5 to 7]

15. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: as for outcome 13
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
units on a scale | 6 [5 to 7] | 6 [5.5 to 7]

16. Secondary Outcome: Functional Ambulation Classification
Description: scored 0 to 5 (non functional ambulator to independant ambulator)
Time Frame: baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 1 [0 to 4] | 1 [0 to 4]

17. Secondary Outcome: Functional Ambulation Classification
Description: scored 0 to 5 (non functional ambulator to independant ambulator)
Time Frame: after treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 1 [0 to 4] | 1 [1 to 4]

18. Secondary Outcome: Functional Ambulation Classification
Description: scored 0 to 5 (non functional ambulator to independant ambulator)
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 1 [0 to 4] | 1 [1 to 4]

19. Secondary Outcome: Walking Ability
Description: The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
Time Frame: baseline
Measure: Median (Full Range); unit: meters
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
meters | 50 [0 to 200] | 60 [1 to 200]

20. Secondary Outcome: Walking Ability
Description: as for outcome 19
Time Frame: after treatment (4th week)
Measure: Median (Full Range); unit: meters
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
meters | 70 [1 to 210] | 70 [5 to 240]

21. Secondary Outcome: Walking Ability
Description: as for outcome 19
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: meters
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
meters | 60 [1 to 210] | 65 [5 to 240]

22. Secondary Outcome: Berg Balance Test (BBT)
Description: Berg Balance Test (BBT) is a functional test with 14 items. Each item is scored on a five point scale (0 to 4) which is determined by ability to perform the task. The total score ranged 0 to 56. A higher score reflects better functional balance.
Time Frame: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 20 [0 to 39] | 15 [5 to 49]

23. Secondary Outcome: Berg Balance Test (BBT)
Description: as for outcome 22
Time Frame: After treatment (4th week)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 24.5 [2 to 42] | 18 [8 to 50]

24. Secondary Outcome: Berg Balance Test (BBT)
Description: as for outcome 22
Time Frame: 3 months after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
Number analyzed (Participants) | 18 | 19
score on a scale | 23 [2 to 40] | 18 [8 to 50]

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Arm/Group | Robot Assisted Training (RAT) | Conventional Training (CT)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03801473/Prot_SAP_000.pdf